CLINICAL TRIAL: NCT05160506
Title: Corticosteroids to Reduce Inflammation in Severe Pancreatitis: A Randomized, Controlled Study
Brief Title: Corticosteroids to Treat Pancreatitis
Acronym: CRISP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P-000803
Record Dates: First submitted 2021-12-07; First posted 2021-12-16 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pancreatitis; Pancreatitis, Acute; Corticosteroid; Hydrocortisone
Keywords: Bedside index of severity in acute pancreatitis; Sequential Organ Failure Assessment; Randomized Controlled Trial
MeSH Terms: conditions — Pancreatitis | interventions — Hydrocortisone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The hydrocortisone and placebo solutions are identical in appearance/volume. Only the research pharmacist, (not a member of either the research or clinical teams) will have access to the treatment allocations to ensure blinding of the investigators and clinical staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydrocortisone (Experimental): Patients in this arm will be administered 100 mg of hydrocortisone in 50 milliliters of saline solution by nursing staff every 8 hours for 72 hours as per standard clinical procedures (9 administrations)
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Patients in this arm will be given matching placebo (50ml 0.9%NACL) by nursing staff every 8 hours for 72 hours (9 administrations)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone is a steroid (corticosteroid) medication.
  Other Names: Cortef; Cortisol; Hydrocort
  Arms: Hydrocortisone
Drug: Placebo — 50ml of 0.9% NACL will serve as the placebo
  Other Names: Normal Saline; 0.9% NACL
  Arms: Placebo

SUMMARY:
This research is being done to determine if the administration of a short course of intravenous hydrocortisone, an anti-inflammatory medication, to patients with severe acute pancreatitis will improve their clinical outcomes and decrease the length of hospitalization. We think that because inflammation in the body drives the progression of pancreatitis, giving a short course of intravenous hydrocortisone may mitigate disease progression and improve clinical outcomes in patients with severe acute pancreatitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study to investigate the effect of intravenous hydrocortisone on clinical outcomes in patients with severe acute pancreatitis. The interventional drug is Hydrocortisone (100 mg of hydrocortisone in 50 milliliters of saline solution). The placebo is saline and is identical in appearance and volume to the interventional drug. Study drug will be administered intravenously every 8 hours for 72 hours as per standard clinical procedures by nursing staff. The patient's sequential organ failure assessment score (SOFA) will be assessed for changes over time. Blood will be drawn at several time points to assess biomarkers over time.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years)
2. Acute pancreatitis as defined by a clinical diagnosis of pancreatitis and a lipase level ≥3x the upper limit of normal.
3. Admission or planned admission to an intensive care unit
4. SOFA disease severity score ≥3 (or at least 3 points above a known baseline)

Exclusion Criteria:

1. Known diagnosis of autoimmune pancreatitis
2. Existing clinical indication for corticosteroids at a dose >5mg of oral prednisone daily (or equivalent)
3. Contraindication to receiving corticosteroids
4. Protected populations (prisoners)
5. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-03-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Severity of Illness Measure | Enrollment to 72 hours
  Change in Sequential Organ failure Assessment (SOFA) Score over 72 hours

SECONDARY OUTCOMES:
Respiratory Failure Measure | Enrollment to 28 days [truncated at 28 days]
  Progression to Acute Respiratory Distress Syndrome (ARDS) assessed as a dichotomous variable for those patients without ARDS upon enrollment
Alive and Ventilator Free Days | Enrollment to 28 days [truncated at 28 days]
  Number of days during the 28-day period after enrollment in which the patient is alive and does not receive mechanical ventilation
Long-term Functional/Quality of Life Measure | 90 days after Enrollment
  Scores from Short Form 36 (SF36), a validated survey used measure health-related quality of life, with higher scores indicating better quality of life.
In-hospital mortality | Enrollment to 90 days [truncated at 90 days]
  Dichotomous variable that assesses whether or not the patient expired prior to hospital discharge
28-day mortality | Enrollment to 28 days [truncated at 28 days]
  Dichotomous variable that indicates whether or not patient expired by the 28-day time-point while enrolled in the trial.
90-day mortality | Enrollment to 90 days [truncated at 90 days]
  Dichotomous variable that indicates whether or not patient expired by the 90-day time-point while enrolled in the trial.
Alive and Hospital free days | Enrollment to 28 days [truncated at 28 days]
  Number of days in which the patient was alive and not in the hospital.
Severity of Illness Measure Stratified By Predicted Survival (Physician Opinion) | Enrollment to 72 hours
  Sequential Organ failure Assessment (SOFA) Score over 72 hours compared for patients stratified by survival likelihood per physician opinion into three subgroups (likely, unlikely, or uncertain)
Severity of Illness Measure Stratified By Bedside Index of Severity in Acute Pancreatitis (BISAP) score | Enrollment to 72 hours
  Sequential Organ failure Assessment (SOFA) Score over 72 hours compared for patients stratified by BISAP scores into two groups (BISAP ≥3; BISAP < 3)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grossestreuer AV, Moskowitz A, Andersen LW, Holmberg MJ, Konacki V, Berg KM, Chase M, Cocchi MN, Donnino MW. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Health-Related Quality of Life in Sepsis. Crit Care Explor. 2020 Nov 23;2(12):e0270. doi: 10.1097/CCE.0000000000000270. eCollection 2020 Dec. PMID 33251516
- [Background] Moskowitz A, Huang DT, Hou PC, Gong J, Doshi PB, Grossestreuer AV, Andersen LW, Ngo L, Sherwin RL, Berg KM, Chase M, Cocchi MN, McCannon JB, Hershey M, Hilewitz A, Korotun M, Becker LB, Otero RM, Uduman J, Sen A, Donnino MW; ACTS Clinical Trial Investigators. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Organ Injury in Septic Shock: The ACTS Randomized Clinical Trial. JAMA. 2020 Aug 18;324(7):642-650. doi: 10.1001/jama.2020.11946. PMID 32809003
- [Background] Donnino MW, Andersen LW, Berg KM, Chase M, Sherwin R, Smithline H, Carney E, Ngo L, Patel PV, Liu X, Cutlip D, Zimetbaum P, Cocchi MN; Collaborating Authors from the Beth Israel Deaconess Medical Center's Center for Resuscitation Science Research Group. Corticosteroid therapy in refractory shock following cardiac arrest: a randomized, double-blind, placebo-controlled, trial. Crit Care. 2016 Apr 3;20:82. doi: 10.1186/s13054-016-1257-x. PMID 27038920
- [Derived] Vine J, Berlin N, Moskowitz A, Berg KM, Liu X, Balaji L, Donnino MW, Grossestreuer AV. Corticosteroids to Reduce Inflammation in Severe Pancreatitis (CRISP) protocol and statistical analysis plan: a prospective, multicentre, double-blind, randomized, placebo controlled clinical trial. Contemp Clin Trials. 2024 Apr;139:107486. doi: 10.1016/j.cct.2024.107486. Epub 2024 Feb 29. PMID 38431131